CLINICAL TRIAL: NCT02769455
Title: Impact of front-of Pack Nutrition Labels on Purchase Intentions in an Online Supermarket-A Series of Randomized Trials
Brief Title: Online Experimental Supermarket
Acronym: SUPERNET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Paris 13 (Other)
Collaborators: Intitut National du Cancer (Unknown)
Responsible Party: Principal Investigator, Serge HERCBERG, Director of Nutritional Epidemiology Research Team, University of Paris 13
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SM2
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Food Selection
Keywords: Food Labelling
MeSH Terms: conditions — Food Preferences | interventions — Recommended Dietary Allowances

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): The control group will not be exposed to any FOP nutrition labels
- Front-of-pack labelling (Reference Intakes) (Experimental): The second group will be exposed to a FOP nutrition label which is already in use on a portion of food products in France: the 'Reference Intakes' (RIs). The RIs are presented in the form of a chain of rectangles presenting the contribution of a portion of the product to a reference balanced diet of an average person (2000kcal) for each of the following nutrients: energy, lipids, saturated fat, sugars and sodium.
  Interventions: Other: Reference intakes
- Front-of-pack labelling (5-CNL) (Experimental): The 5-CNL was developed as a colour-coded summary system nutrition label, following the elements pointed out in reviews.
  The format of the 5-CNL system therefore includes five categories of nutritional quality of food products, ranging from green (Associated with the A grade) for foods of the highest nutritional quality to red (associated with the E grade), for products with lower nutritional quality. The format is presented in the form of a continuous chain of rectangles, each with its own letter/colour, the letter/colour corresponding to the product being enlarged.
  Interventions: Other: 5-CNL

INTERVENTIONS:
Other: Reference intakes — FOP nutrition label which is already in use on a portion of food products in France: the 'Reference Intakes' (RIs). The RIs are a chain of rectangles presenting the contribution of a portion of the product to a reference balanced diet of an average person (2000kcal) for each of the following nutrients: energy, lipids, saturated fat, sugars and sodium.
  The presentation of the products will always include the label affixed on it. Moreover, the product pages will include two pictures of the product: one with only the package (including the RI as FOP labelling), and a picture with both the package and a larger version of the label, so that it is more visible to the participant. These elements ensure higher visibility, awareness and understanding of the label.
  Arms: Front-of-pack labelling (Reference Intakes)
Other: 5-CNL — The 5-CNL was developed as a colour-coded summary system nutrition label, following the elements pointed out in reviews.
  The format includes five categories, ranging from green (Associated with the A grade) for foods of the highest nutritional quality to red (associated with the E grade), for products with lower nutritional quality. The format is presented in the form of a continuous chain of rectangles, each with its own letter/colour, the one corresponding to the product being enlarged.
  The presentation of the products will always include the label affixed on it. Two pictures of the product will be included: one with only the package (including the 5-CNL as FOP labelling), and a picture with both the package and a larger version of the label, so that it is more visible to the participant.
  Arms: Front-of-pack labelling (5-CNL)

SUMMARY:
Front-Of-Pack (FOP) nutrition labelling, providing simplified information on nutritional content at a glance, in order to help consumer make informed choices, has been identified as of major interest by public health specialists of many countries. French health authorities are currently considering the endorsement of a FOP nutrition label, but no specific format has yet been determined. A more simplified FOP nutrition label has been put forward in France, the 5-Colour Nutrition Label (5-CNL). Recent data suggests that the 5-CNL FOP label is well perceived and understood by consumers. The introduction of a FOP nutrition labelling system has been identified as challenging in certain population groups, due to their lower level of nutrition knowledge and unhealthier diets.

The aim of the investigators is to evaluate the impact of FOP nutrition labels on the nutritional quality of the shopping cart in an online experimental supermarket in various nutritionally at-risk populations. Two FOP systems will be tested to a control situation without FOP labelling: the Reference Intakes (RI), currently in use by some manufacturers and present in a portion of food products sold in France, and the 5-Colour Nutrition Label (5-CNL).

Three 3 arm parallel arm randomized trials are designed, each targeting a specific population. The methodology and interventions are identical across trials. Trials will be conducted in: 1) Working adults between 30-50 years old with low income, 2) Students and 3) Older subjects with identified chronic diseases. The intervention consists in the application of FOP nutrition labels on all food products, either the RI label, currently in use in some products in France, and the 5-CNL label. A control situation with no FOP will also be used. Participants will be asked to perform a shopping session in an experimental online supermarket, in one of the three experimental conditions described. The main outcome will be the overall nutritional quality of the shopping cart, assessed using the mean Food Standards Agency Nutrient profiling system score of the items in the shopping cart.

DETAILED DESCRIPTION:
Front-Of-Pack (FOP) nutrition labelling, providing simplified information on nutritional content at a glance, in order to help consumer make informed choices, has been identified as of major interest by public health specialists of many countries. Modelling studies suggested that adoption of effective nutrition labelling would be cost-effective and provide health benefits. French health authorities are currently considering the endorsement of a FOP nutrition label, but no specific format has yet been determined. A more simplified FOP nutrition label has been put forward in France, the 5-Colour Nutrition Label (5-CNL). Recent data suggests that the 5-CNL FOP label is well perceived and understood by consumers. Moreover, a recent randomized trial, based on an online experimental supermarket, showed that the 5-CNL displayed the highest difference in nutritional quality compared to the control situation. The introduction of a FOP nutrition labelling system has been identified as challenging in certain population groups, due to their lower level of nutrition knowledge and unhealthier diets. Subjects with lower levels of income, or the young appear as a key target in which the impact of FOP nutrition labels has been poorly explored. Moreover, the impact of such a label on subjects suffering from a chronic condition for which dietary modifications are part of the treatment should be carefully considered, in order to avoid potential undesirable effects of the label in these populations.

The aim of the investigators is to evaluate the impact of FOP nutrition labels on the nutritional quality of the shopping cart in an online experimental supermarket in various nutritionally at-risk populations. Two FOP systems will be tested to a control situation without FOP labelling: the Reference Intakes (RI), currently in use by some manufacturers and present in a portion of food products sold in France, and the 5-Colour Nutrition Label (5-CNL).

Three 3 arm parallel arm randomized trials are designed, each targeting a specific population. The methodology and interventions are identical across trials. Trials will be conducted in: 1) Working adults between 30-50 years old with low income, 2) Students and 3) Older subjects with identified chronic diseases. The intervention consists in the application of FOP nutrition labels on all food products, either the RI label, currently in use in some products in France, and the 5-CNL label. A control situation with no FOP will also be used. Participants will be asked to perform a shopping session in an experimental online supermarket, in one of the three experimental conditions described. The main outcome will be the overall nutritional quality of the shopping cart, assessed using the mean Food Standards Agency Nutrient profiling system score of the items in the shopping cart.

ELIGIBILITY:
TRIAL n°1

Inclusion Criteria:

* Subjects 30-50 years old
* Having finished their studies and currently active (either working or unemployed)
* Income/UC <1200€/month

Exclusion Criteria:

* Student, retired
* Subjects living outside of mainland France
* Subjects never engaging in grocery shopping

TRIAL N°2

Inclusion Criteria:

* Subject 18-25 years old
* Self-declared as student

Exclusion Criteria:

• Subjects never engaging in grocery shopping

TRIAL N°3

Inclusion Criteria:

* Subjects >50 years-old
* Diagnosed with one or more of the following chronic conditions (self-reported) : type 2 diabetes, dislipidemia (elevated cholesterol levels, low HDL cholesterol levels, elevated triglycerides levels), hypertension, cardiovascular disease, obesity

Exclusion Criteria:

* Subjects declaring suffering from none of the mentioned chronic conditions
* Subjects never engaging in grocery shopping

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
FSA Score | 3 months
  Mean nutritional quality of the items in the shopping cart, using the mean Food Standards Agency nutrient profiling system (FSA score) of the items in the shopping cart. The FSA score for foods and beverages is computed taking into account nutrient content for 100g. It allocates positive points (0-10) for content in energy (KJ), total sugar (g), saturated fatty acids (g) and sodium (mg). Negative points (0-5) are allocated to content in fruits, vegetables, legumes and nuts (%), fibers (g) and proteins (g). Scores for foods and beverages were therefore based on a discrete continuous scale from -15 (most healthy) to +40 (less healthy). Modifications to the original score were used in order to ensure a higher consistency with French nutritional recommendations for beverages, cheese and added fats

SECONDARY OUTCOMES:
Calories (/100g) | 3 months
  Mean calorie density of the items in the shopping cart. Calorie content per 100g for each item is taken into account. No weighing on total energy or weight of the shopping cart.
Saturates (g/100g) | 3 months
  Mean saturated fat content of the items in the shopping cart. Saturates content per 100g for each item is taken into account. No weighing on total energy or weight of the shopping cart.
Sugar (g/100g) | 3 months
  Mean sugar content of the items in the shopping cart. Sugar content per 100g for each item is taken into account. No weighing on total energy or weight of the shopping cart.
Sodium (mg/100g) | 3 months
  Mean sodium content of the items in the shopping cart. Sodium content per 100g for each item is taken into account. No weighing on total energy or weight of the shopping cart.
Fibers (g/100g) | 3 months
  Mean fiber content of the items in the shopping cart. Fiber content per 100g for each item is taken into account. No weighing on total energy or weight of the shopping cart.
Proteins (g/100g) | 3 months
  Mean protein content of the items in the shopping cart. Protein content per 100g for each item is taken into account. No weighing on total energy or weight of the shopping cart.
Fruits and vegetables (%/100g) | 3 months
  Mean fruit and vegetables content of the items in the shopping cart. Fruits and vegetables content per 100g for each item is taken into account. No weighing on total energy or weight of the shopping cart.

CONTACTS AND LOCATIONS:
Overall Officials: Serge Hercberg, Principal Investigator — Nutritional Epidemiology Research Team
Locations (1):
- Equipe de Recherche en Epidémiologie Nutritionnelle, Bobigny, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Egnell M, Boutron I, Peneau S, Ducrot P, Touvier M, Galan P, Fezeu L, Porcher R, Ravaud P, Hercberg S, Kesse-Guyot E, Julia C. Impact of the Nutri-Score front-of-pack nutrition label on purchasing intentions of individuals with chronic diseases: results of a randomised trial. BMJ Open. 2022 Aug 29;12(8):e058139. doi: 10.1136/bmjopen-2021-058139. PMID 36038180
- [Derived] Egnell M, Galan P, Fialon M, Touvier M, Peneau S, Kesse-Guyot E, Hercberg S, Julia C. The impact of the Nutri-Score front-of-pack nutrition label on purchasing intentions of unprocessed and processed foods: post-hoc analyses from three randomized controlled trials. Int J Behav Nutr Phys Act. 2021 Mar 17;18(1):38. doi: 10.1186/s12966-021-01108-9. PMID 33731145
- [Derived] Egnell M, Boutron I, Peneau S, Ducrot P, Touvier M, Galan P, Buscail C, Porcher R, Ravaud P, Hercberg S, Kesse-Guyot E, Julia C. Randomised controlled trial in an experimental online supermarket testing the effects of front-of-pack nutrition labelling on food purchasing intentions in a low-income population. BMJ Open. 2021 Feb 8;11(2):e041196. doi: 10.1136/bmjopen-2020-041196. PMID 33558350